CLINICAL TRIAL: NCT01332981
Title: Overall Survival Estimation After a 7 Year Follow-up in Metastatic Breast Cancer Patients Treated by Herceptin® as 1st Line Therapy (Post-HERMINE Study)
Brief Title: An Observational Follow-up Study of 1st-Line Treatment With Herceptin (Trastuzumab) in Patients With Metastatic Breast Cancer (Post-HERMINE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22958
Record Dates: First submitted 2011-04-06; First posted 2011-04-11 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This is an observational follow-up study on the efficacy of 1st-line treatment with Herceptin (trastuzumab) in patients with metastatic breast cancer 7 years after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patient, >/= 18 years of age
* Metastatic breast cancer
* 1st-line treatment with Herceptin initiated in 2002
* Included in pharmaco-epidemiologic HERMINE study

Exclusion Criteria:

* Patient died before scheduled follow-up visit (March 2005)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast cancer patients treated by Herceptin® as 1st line therapy
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This post-HERMINE study was an observational, pharmaco-epidemiological, and retrospective study. Among the 102 participants who were alive at the end of the observation period in the HERMINE study, 69 were included in the post-HERMINE study from 31 centers in France. The study was conducted between 23 February 2010 to 15 October 2010.
Pre-assignment Details: Overall analysis population was 220. During data check for the participants alive at the end of HERMINE study, it appeared that 1 participant was included twice. Thus, the real no. that started treatment with 1st-line trastuzumab therapy was 220 and not 221. Thus, the no. of participants still alive at the end of HERMINE study was 102 and not 103.
Groups:
- Trastuzumab: Female participants with overexpression of human epidermal growth factor receptor 2 (HER2+) metastatic breast cancer treated with trastuzumab as first-line treatment since 2002, included in the pharmaco-epidemiological HERMINE study and were still alive at the end of the observation period in March 2005.
Period: Overall Study
Arm/Group | Trastuzumab
Started | 220
Completed | 220
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis population included participants with HER2+ metastatic breast cancer included in HERMINE study and treated with trastuzumab as first line therapy.
Groups:
- Transtuzumab: Female participants with overexpression of human epidermal growth factor receptor 2 (HER2+) metastatic breast cancer treated with trastuzumab as first-line treatment since 2002, included in the pharmaco-epidemiological HERMINE study and were still alive at the end of the observation period in March 2005.
Arm/Group | Transtuzumab
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: The time between the first infusion of trastuzumab and the date of death from any cause. Participants who were still alive at the end of the post-HERMINE study or lost to follow-up were censored at the last date they were known to be alive.
Time Frame: Up to 7 years
Population: Participants with HER2+ metastatic breast cancer included in HERMINE study and treated with trastuzumab as first line therapy.
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Transtuzumab
Number analyzed (Participants) | 220
Years | 2.51 [2.02 to 3.02]

2. Secondary Outcome: Median Time to Progression-Free Survival
Description: The Progression-Free Survival (PFS) was defined as the time between the treatment start date (date of the first trastuzumab infusion) and the date of the first disease progression or disease-related death. Participants who had not progressed at the end of the post-HERMINE study were censored at the last date they were known to be alive. Progression-Free Survival was estimated by using Kaplan-Meier method.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Transtuzumab
Number analyzed (Participants) | 220
Years | 0.85 [0.76 to 1.03]

3. Secondary Outcome: Median Time to Progression
Description: The Time to Progression (TTP) was defined as the time between the treatment start date (date of the first trastuzumab infusion) and the date of the first disease progression or disease-related death. Participants who had not progressed at the end of the post-HERMINE study were censored at the last date they were known to be alive. If the cause of death was unknown, the death was considered for this analysis as due to the disease. All participants who did not progress, the death was considered to be due to the disease.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Transtuzumab
Number analyzed (Participants) | 220
Years | 0.85 [0.76 to 1.03]

4. Secondary Outcome: Median Treatment Duration and the Duration of Exposure to Trastuzumab
Description: Treatment duration was defined as the time between the first and the last infusion of trastuzumab. Exposure duration was defined only for the participants who continued trastuzumab after HERMINE study, as the sum of treatment duration as part of HERMINE study and of the treatment durations as part of post-HERMINE study taking into account temporary treatment discontinuations. For analyses of treatment and exposure duration , dates of infusion of trastuzumab were missing for 18 participants, so treatment and exposure durations were calculated for only 202 participants.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Median (Full Range); unit: Years
Arm/Group | Trastuzumab
Number analyzed (Participants) | 220
Years
  Total treatment duration, n=202 | 1.19 [0.00 to 8.68]
  Exposure duration, n=202 | 3.98 [1.04 to 8.06]

5. Secondary Outcome: Prognostic Factors for Overall Survival
Description: Search for prognostic factors for OS was performed using Cox regression model. First, all parameters were analyzed in univariate models, and the hypothesis of proportional risks was tested. Significant parameters at 15%-level were retained for the multivariate model. For the multivariate analysis, two models were built for prognostic factors for OS. In the first one (Model 1), a stepwise selection method was used on all parameters that were significant in the univariate analyses, whatever the significance level of the associations between parameters. In the second one (Model 2), a stepwise selection was used on the significant parameters that were not correlated. The significance level for entry was 10% and the significance level for removal was 5%. The variables n°5 and n°6 were found to be significantly associated, thus only the variable n°6 was tested in the Model 2. This variable was not retained by the stepwise selection in the Model 1, contrary to the variable n°5.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Groups:
- Model 1: In the first one (Model 1), a stepwise selection method was used on all parameters that were significant in the univariate analyses, whatever the significance level of the associations between parameters.
- Model 2: In the second one (Model 2), a stepwise selection was used on the significant parameters that were not correlated. The significance level for entry was 10% and the significance level for removal was 5%.
Arm/Group | Model 1 | Model 2
Number analyzed (Participants) | 220 | 220
Hazard Ratio
  Scarff-Bloom-Richardson grade, increase >1 | 1.55 [1.10 to 2.19] | 1.49 [1.06 to 2.08]
  Liver metastases at beginning of treatment, Yes/No | 1.60 [1.12 to 2.28] | 1.55 [1.10 to 2.19]
  CNS metastases at begining of treatment, Yes/No | 4.63 [2.36 to 9.09] | 4.70 [2.40 to 9.20]
  Time of first metastases and dose (mnths), >1 mnth | 1.04 [1.01 to 1.06] | 1.04 [1.01 to 1.06]
  Time:Diagnosis and 1st metastic relapse <=/>=2 Yrs | 0.52 [0.36 to 0.75] | NA [NA to NA] — The variables n°5 and n°6 were found to be significantly associated, thus only the variable n°6 was tested in the Model 2. This variable was not retained by the stepwise selection in the Model 1, contrary to the variable n°5.
  Time:Diagnosis and 1st metastic relapse <=/>=24 m | NA [NA to NA] — The variables n°5 and n°6 were found to be significantly associated, thus only the variable n°6 was tested in the Model 2. This variable was not retained by the stepwise selection in the Model 1, contrary to the variable n°5. | 0.54 [0.38 to 0.78]

6. Secondary Outcome: Prognostic Factors For Time to Progression
Description: Prognostic factors for TTP were searched by using Cox regression model. First, all parameters were analysed in univariate models, and the hypothesis of proportional risks was tested. Significant parameters at 15% level were retained for multivariate model. For multivariate analyses, 2 models were built for prognostic factor of TTP. In Model 1, stepwise selection method was used on all parameters that were significant in the univariate analyses, whatever the significance level of the associations between parameters. In Model 2, stepwise selection was used on the significant parameters that were not correlated. The significance level for entry was 10% and the significance level for exit was 5%. Six parameters remained in the Model 1 to search for prognostic factors of TTP. Once the correlated variables were removed, there were only 3 variables left in Model 2: the age was not kept by the stepwise selection. Results below are for Model 1 and similar results were obtained for Model 2
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Model 1 | Model 2
Number analyzed (Participants) | 220 | 220
Hazard Ratio
  No.of metastatic sites at trtmnt start,1/2/>2, >1 | 1.34 [1.10 to 1.62] | NA [NA to NA] — Six parameters remained in the Model 1 to search for prognostic factors of TTP. Once the correlated variables were removed, there were only three variables left in Model 2: the age was not kept by the stepwise selection.
  Liver metastases at start of the treatment Yes/No | 1.44 [1.06 to 1.94] | 1.48 [1.10 to 1.98]
  CNS metastases at start of the treatment Yes/No | 2.81 [1.51 to 5.22] | 3.94 [2.18 to 7.10]
  Time of first metastases and dose (mnths), >1 mnth | 1.03 [1.01 to 1.06] | NA [NA to NA] — Six parameters remained in the Model 1 to search for prognostic factors of TTP. Once the correlated variables were removed, there were only three variables left in Model 2: the age was not kept by the stepwise selection.
  Age in class ≥50 years old / <50 years old | 0.69 [0.50 to 0.94] | NA [NA to NA] — Six parameters remained in the Model 1 to search for prognostic factors of TTP. Once the correlated variables were removed, there were only three variables left in Model 2: the age was not kept by the stepwise selection.
  Time:Diagnosis and 1st metastic relapse <=/>=2 Yrs | 0.64 [0.47 to 0.86] | 0.68 [0.50 to 0.91]

ADVERSE EVENTS:
Time Frame: Up to 7 Years
Description: This observational retrospective study was conducted to provide an update to the OS of participants with metastatic breast cancer, 7 years after starting first-line treatment with trastuzumab in subgroup of participants included in HERMINE study. Therefore, serious adverse event and non-serious adverse event data were not collected in this study.
Arm/Group | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.